CLINICAL TRIAL: NCT01440413
Title: Study of the Response to a Neoadjuvant Chemotherapy Based on the Antitumor Immune Response in Localized Breast Cancer
Acronym: BREAST IMMUN
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Centre Leon Berard (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: BREAST IMMUN; ET11-059 (Other: Sponsor identification)
Record Dates: First submitted 2011-09-14; First posted 2011-09-26 (Estimated); Last update posted 2020-03-24 (Actual); Status verified 2020-03

CONDITIONS: Breast Cancer
Keywords: anti-tumor immune response; neo-adjuvant chemotherapy; relapse; long term survival; histo-pathological response; tumor cell death; tumor associated antigens; Calreticulin; Localized breast cancer
MeSH Terms: conditions — Breast Neoplasms; Recurrence | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Biological: Blood and tumor sample — Blood samples will be collected on the first day of the first cycle of chemotherapy (before injection of chemotherapy), on the first day of the third cycle (before injection of chemotherapy), on day of surgery and 6 months after surgery and in case of relapse.
  Tumor samples will be collected on diagnosis, on surgery and on the first day of the third chemotherapy course (optional).

SUMMARY:
This is a prospective, non-randomized study which aims to evaluate the response to a neoadjuvant chemotherapy according to the the antitumor immune response in localized breast cancer.

40 patients will be enrolled in the study. They will receive chemotherapy : 3 or 4 anthracycline cycles or 3 or 4 FEC-100 cycles followed by 3 or 4 taxane cycles.

Trastuzumab will be added to taxane for HER2+/Neu+ patients. Then, patients will be operated and receive an adjuvant treatment which will both depend on the investigator's appreciation.

Blood sample will be collected on the first day of the first chemotherapy cycle, on the first day of the third cycle, on surgery, 6 months after the surgery and in case of relapse.

Tumor sample will be collected on diagnosis as much as possible and on surgery.

Patients will be followed during 5 years.

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven localized breast cancer required anthracycline chemotherapy +/- trastuzumab before surgery
* Age > 18 years
* Chemotherapy with 3 anthracycline cycles to begin (doxorubicin or epirubicin)
* Any previous treatment for this cancer
* Performance Status <= 1
* Agreement for the conservation of biological samples
* Covered by an medical insurance
* Signed written informed consent form
* Availability of tumoral sample collected at diagnosis

Exclusion Criteria:

* Previous surgery for the breast cancer
* Already under chemotherapy before the first blood sample
* Previous Antitumoral treatment
* Under immunosuppressive treatment
* Under corticoids during the 15 days before enrollment
* History of concomitant cancer except if it has been cured for at least 5 years
* History of lymphoma or breast sarcoma
* History of chronic inflammatory disease or autoimmune disease, hepatitis B or C or immune dysfunction disease (including HIV-positive stage AIDS) known
* History of other disease which is discrepant with this study
* Deprived of liberty by court or administrative decision
* Pregnant or breastfeeding women or with no use of effective birth control methods for women of childbearing potential

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2011-12 (Actual); Primary Completion 2018-12 (Actual); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Determine the correlation between histopathological response (pCR) and induction of tumor immunity in response to neoadjuvant chemotherapy | Day (D) 1 chemotherapy (CT) n°1, D1 CT n°3, Surgery, 6 month post surgery
  Rate of histopathologic response (IHC). Analysis of lymphocyte subpopulations (whole blood - flow cytometry). Analysis of the frequency of immune cells, the phenotype and functional status on the site of the tumor (fixed tissue - IHC). Analysis of the functional status of sub-populations of DC and lymphocytes of innate immunity (fresh whole blood - flow cytometry). Analysis of BCR and TCR repertoires (mononuclear cells - PCR). Identification of TAA expressed by the tumor (plasma, tumor - ELISA, IHC).Analysis of the humoral response against TAA (plasma - ELISA).

SECONDARY OUTCOMES:
Evolution of the immune profile during management of localized breast cancer | D1 CT n°1, D1 CT n°3, Surgery, 6 month post surgery
  Analysis in plasma of the rate of apoptotic tumor cells, of TAA (CEA and MUC1 ELISA), of tumor DNA and endogenous ligands of TLR (HMGB1 ELISA) Assay of cytokines and chemokines in plasma Analysis of the expression of proteins involved in the translocation of CRT to the cell surface (fixed-frozen tissue - IHC or immunoblotting) Analysis on the tumor (IHC or immunoblotting) of degradation of BAP31, activation of caspase 8/Bax/Bak, phosphorylation of eIF2 and exposure of surface CRT, KDEL receptor and ERp57
Analysis of genetic polymorphisms | D1 CT n°1, D1 CT n°3, Surgery, 6 month post surgery
  Analysis of P2X7 and TLR4 polymorphisms on circulating cells (plasma)
Determination of relapse risk based on biological characteristics identified | At the end of the study (5 years of follow-up)
  Progression-free survival
Determining the risk of death based on biological characteristics identified | At the end of the study (5 years of follow-up)
  Overall survival

CONTACTS AND LOCATIONS:
Overall Officials: Olivier TREDAN, MD, Principal Investigator — Centre Leon Berard
Locations (2):
- France (2):
  - Centre Georges François Leclerc, Dijon
  - Centre Leon Berard, Lyon

REFERENCES:
- [Background] Apetoh L, Ghiringhelli F, Tesniere A, Obeid M, Ortiz C, Criollo A, Mignot G, Maiuri MC, Ullrich E, Saulnier P, Yang H, Amigorena S, Ryffel B, Barrat FJ, Saftig P, Levi F, Lidereau R, Nogues C, Mira JP, Chompret A, Joulin V, Clavel-Chapelon F, Bourhis J, Andre F, Delaloge S, Tursz T, Kroemer G, Zitvogel L. Toll-like receptor 4-dependent contribution of the immune system to anticancer chemotherapy and radiotherapy. Nat Med. 2007 Sep;13(9):1050-9. doi: 10.1038/nm1622. Epub 2007 Aug 19. PMID 17704786
- [Background] Banchereau J, Briere F, Caux C, Davoust J, Lebecque S, Liu YJ, Pulendran B, Palucka K. Immunobiology of dendritic cells. Annu Rev Immunol. 2000;18:767-811. doi: 10.1146/annurev.immunol.18.1.767. PMID 10837075
- [Background] Bates GJ, Fox SB, Han C, Leek RD, Garcia JF, Harris AL, Banham AH. Quantification of regulatory T cells enables the identification of high-risk breast cancer patients and those at risk of late relapse. J Clin Oncol. 2006 Dec 1;24(34):5373-80. doi: 10.1200/JCO.2006.05.9584. PMID 17135638
- [Background] Bear HD, Anderson S, Smith RE, Geyer CE Jr, Mamounas EP, Fisher B, Brown AM, Robidoux A, Margolese R, Kahlenberg MS, Paik S, Soran A, Wickerham DL, Wolmark N. Sequential preoperative or postoperative docetaxel added to preoperative doxorubicin plus cyclophosphamide for operable breast cancer:National Surgical Adjuvant Breast and Bowel Project Protocol B-27. J Clin Oncol. 2006 May 1;24(13):2019-27. doi: 10.1200/JCO.2005.04.1665. Epub 2006 Apr 10. PMID 16606972
- [Background] Blay JY, Chauvin F, Le Cesne A, Anglaret B, Bouhour D, Lasset C, Freyer G, Philip T, Biron P. Early lymphopenia after cytotoxic chemotherapy as a risk factor for febrile neutropenia. J Clin Oncol. 1996 Feb;14(2):636-43. doi: 10.1200/JCO.1996.14.2.636. PMID 8636781
- [Background] Borg C, Ray-Coquard I, Philip I, Clapisson G, Bendriss-Vermare N, Menetrier-Caux C, Sebban C, Biron P, Blay JY. CD4 lymphopenia as a risk factor for febrile neutropenia and early death after cytotoxic chemotherapy in adult patients with cancer. Cancer. 2004 Dec 1;101(11):2675-80. doi: 10.1002/cncr.20688. PMID 15503313
- [Background] Chapman C, Murray A, Chakrabarti J, Thorpe A, Woolston C, Sahin U, Barnes A, Robertson J. Autoantibodies in breast cancer: their use as an aid to early diagnosis. Ann Oncol. 2007 May;18(5):868-73. doi: 10.1093/annonc/mdm007. Epub 2007 Mar 7. PMID 17347129
- [Background] Disis ML, Knutson KL, Schiffman K, Rinn K, McNeel DG. Pre-existent immunity to the HER-2/neu oncogenic protein in patients with HER-2/neu overexpressing breast and ovarian cancer. Breast Cancer Res Treat. 2000 Aug;62(3):245-52. doi: 10.1023/a:1006438507898. PMID 11072789
- [Background] Domschke C, Schuetz F, Ge Y, Seibel T, Falk C, Brors B, Vlodavsky I, Sommerfeldt N, Sinn HP, Kuhnle MC, Schneeweiss A, Scharf A, Sohn C, Schirrmacher V, Moldenhauer G, Momburg F, Beckhove P. Intratumoral cytokines and tumor cell biology determine spontaneous breast cancer-specific immune responses and their correlation to prognosis. Cancer Res. 2009 Nov 1;69(21):8420-8. doi: 10.1158/0008-5472.CAN-09-1627. Epub 2009 Oct 20. PMID 19843863
- [Background] Fan C, Oh DS, Wessels L, Weigelt B, Nuyten DS, Nobel AB, van't Veer LJ, Perou CM. Concordance among gene-expression-based predictors for breast cancer. N Engl J Med. 2006 Aug 10;355(6):560-9. doi: 10.1056/NEJMoa052933. PMID 16899776
- [Background] Guckel B, Rentzsch C, Nastke MD, Marme A, Gruber I, Stevanovic S, Kayser S, Wallwiener D. Pre-existing T-cell immunity against mucin-1 in breast cancer patients and healthy volunteers. J Cancer Res Clin Oncol. 2006 Apr;132(4):265-74. doi: 10.1007/s00432-005-0064-6. Epub 2005 Dec 22. PMID 16374613
- [Background] Loprinzi CL, Thome SD. Understanding the utility of adjuvant systemic therapy for primary breast cancer. J Clin Oncol. 2001 Feb 15;19(4):972-9. doi: 10.1200/JCO.2001.19.4.972. PMID 11181659
- [Background] Ray-Coquard I, Ghesquiere H, Bachelot T, Borg C, Biron P, Sebban C, LeCesne A, Chauvin F, Blay JY; ELYPSE Study Group. Identification of patients at risk for early death after conventional chemotherapy in solid tumours and lymphomas. Br J Cancer. 2001 Sep 14;85(6):816-22. doi: 10.1054/bjoc.2001.2011. PMID 11556830
- [Background] Remontet L, Esteve J, Bouvier AM, Grosclaude P, Launoy G, Menegoz F, Exbrayat C, Tretare B, Carli PM, Guizard AV, Troussard X, Bercelli P, Colonna M, Halna JM, Hedelin G, Mace-Lesec'h J, Peng J, Buemi A, Velten M, Jougla E, Arveux P, Le Bodic L, Michel E, Sauvage M, Schvartz C, Faivre J. Cancer incidence and mortality in France over the period 1978-2000. Rev Epidemiol Sante Publique. 2003 Feb;51(1 Pt 1):3-30. PMID 12684578
- [Background] Rentzsch C, Kayser S, Stumm S, Watermann I, Walter S, Stevanovic S, Wallwiener D, Guckel B. Evaluation of pre-existent immunity in patients with primary breast cancer: molecular and cellular assays to quantify antigen-specific T lymphocytes in peripheral blood mononuclear cells. Clin Cancer Res. 2003 Oct 1;9(12):4376-86. PMID 14555509
- [Background] Rosenberg SA. Shedding light on immunotherapy for cancer. N Engl J Med. 2004 Apr 1;350(14):1461-3. doi: 10.1056/NEJMcibr045001. No abstract available. PMID 15070799
- [Background] Sakaguchi S. Naturally arising CD4+ regulatory t cells for immunologic self-tolerance and negative control of immune responses. Annu Rev Immunol. 2004;22:531-62. doi: 10.1146/annurev.immunol.21.120601.141122. PMID 15032588
- [Background] Thomachot MC, Bendriss-Vermare N, Massacrier C, Biota C, Treilleux I, Goddard S, Caux C, Bachelot T, Blay JY, Menetrier-Caux C. Breast carcinoma cells promote the differentiation of CD34+ progenitors towards 2 different subpopulations of dendritic cells with CD1a(high)CD86(-)Langerin- and CD1a(+)CD86(+)Langerin+ phenotypes. Int J Cancer. 2004 Jul 10;110(5):710-20. doi: 10.1002/ijc.20146. PMID 15146561
- [Background] Treilleux I, Blay JY, Bendriss-Vermare N, Ray-Coquard I, Bachelot T, Guastalla JP, Bremond A, Goddard S, Pin JJ, Barthelemy-Dubois C, Lebecque S. Dendritic cell infiltration and prognosis of early stage breast cancer. Clin Cancer Res. 2004 Nov 15;10(22):7466-74. doi: 10.1158/1078-0432.CCR-04-0684. PMID 15569976
- [Background] van 't Veer LJ, Dai H, van de Vijver MJ, He YD, Hart AA, Mao M, Peterse HL, van der Kooy K, Marton MJ, Witteveen AT, Schreiber GJ, Kerkhoven RM, Roberts C, Linsley PS, Bernards R, Friend SH. Gene expression profiling predicts clinical outcome of breast cancer. Nature. 2002 Jan 31;415(6871):530-6. doi: 10.1038/415530a. PMID 11823860
- [Background] van de Vijver MJ, He YD, van't Veer LJ, Dai H, Hart AA, Voskuil DW, Schreiber GJ, Peterse JL, Roberts C, Marton MJ, Parrish M, Atsma D, Witteveen A, Glas A, Delahaye L, van der Velde T, Bartelink H, Rodenhuis S, Rutgers ET, Friend SH, Bernards R. A gene-expression signature as a predictor of survival in breast cancer. N Engl J Med. 2002 Dec 19;347(25):1999-2009. doi: 10.1056/NEJMoa021967. PMID 12490681
- [Background] Zitvogel L, Tesniere A, Kroemer G. Cancer despite immunosurveillance: immunoselection and immunosubversion. Nat Rev Immunol. 2006 Oct;6(10):715-27. doi: 10.1038/nri1936. Epub 2006 Sep 15. PMID 16977338
- [Background] Zou W. Immunosuppressive networks in the tumour environment and their therapeutic relevance. Nat Rev Cancer. 2005 Apr;5(4):263-74. doi: 10.1038/nrc1586. PMID 15776005
- [Background] Obeid M, Tesniere A, Ghiringhelli F, Fimia GM, Apetoh L, Perfettini JL, Castedo M, Mignot G, Panaretakis T, Casares N, Metivier D, Larochette N, van Endert P, Ciccosanti F, Piacentini M, Zitvogel L, Kroemer G. Calreticulin exposure dictates the immunogenicity of cancer cell death. Nat Med. 2007 Jan;13(1):54-61. doi: 10.1038/nm1523. Epub 2006 Dec 24. PMID 17187072